CLINICAL TRIAL: NCT02451826
Title: A Randomized Study to Evaluate the Effect of a Contraceptive Vaginal Ring Delivering a Daily Dose of 2500 μg of Ulipristal Acetate Combined With a Single or Repeated Levonorgestrel 1.5mg Oral Dose on Inhibition of Ovulation, Endometrial Changes and Bleeding Patterns in Normal Cycling Women
Brief Title: A Study to Evaluate the Effect of a Contraceptive Vaginal Ring Delivering Ulipristal Acetate Combined With a Single or Repeated Levonorgestrel on Inhibition of Ovulation, Endometrial Changes and Bleeding Patterns in Normal Cycling Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 674
Record Dates: First submitted 2015-04-16; First posted 2015-05-22 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Ovulation Inhibition
Keywords: ovulation inhibition; endometrial changes; bleeding patterns
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.5 mg tablet LNG after 12 weeks (Active Comparator): CVR delivering 2,500 µg of Ulipristal acetate per day and a single dose of levonorgestrel delivered in a 1.5 mg tablet after 12 weeks of CVR use
  Interventions: Drug: Ulipristal acetate
- 1.5 mg tablet LNG every 4 weeks (Active Comparator): CVR delivering 2,500 µg of Ulipristal acetate per day and one 1.5 mg tablet levonorgestrel every 4 weeks of CVR use (three times).
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — CVR delivering Ulipristal acetate and one tablet levonorgestrel.

SUMMARY:
The purpose of this study is to determine the effect of a contraceptive vaginal ring on inhibition of ovulation, endometrial changes and bleeding patterns in normal cycling women.

ELIGIBILITY:
Inclusion Criteria:

* Not at risk for pregnancy based on one of the following: a. subject has undergone sterilization; b. subject is monogamous and her male partner has undergone sterilization
* Have regular menstrual cycles of 25-35 days duration
* Have an intact uterus and both ovaries
* Will be able to comply with the protocol
* Capable of giving informed consent

Exclusion Criteria:

* Women participating in another clinical trial
* Women not living in the catchment area of the clinic
* Known hypersensitivity to progestins or antiprogestins
* Known hypersensitivity to silicone rubber
* Any chronic disease
* All contraindications to oral contraceptive use, including: a. Thrombophlebitis or thromboembolic disorders; b. Past history of deep vein thrombophlebitis or thromboembolic disorders; c. Past or current cerebrovascular or coronary artery disease; d. Migraine with focal aura; e. Known or suspected carcinoma of the breast; f. Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia; g. Undiagnosed abnormal genital bleeding; h. Cholestatic jaundice of pregnancy or jaundice with prior pill use; i. Hepatic adenomas or carcinomas; j. Known or suspected pregnancy
* Desire to get pregnant during the study (through the use of reproductive technology for sterilized women or vasectomy reversal for sterilized partners)
* Breastfeeding
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities
* Women with a current abnormal Pap: In accordance with the Bethesda system of classification: smear suggestive of high-grade pre-cancerous lesion(s), including HGSIL, are excluded; Women with LGSIL or ASCUS/high-risk HPV positive may participate if further evaluated with colposcopy and biopsy and no evidence of a lesion with a severity > CIN I is present and/or endocervical curettage is negative; Women with a biopsy finding of CIN I should have follow up for this finding per standard of care; women are excluded it treatment is indicated.
* Known benign or malignant liver tumors; known active liver disease
* Cancer (past history of any carcinoma or sarcoma)
* Medically diagnosed severe depression currently or in the past
* Known or suspected alcoholism or drug abuse
* Abnormal serum fasting clinical chemistry values
* Women with known abnormal thyroid status
* Women with known impaired hypothalamic-pituitary-adrenal reserve
* Average diastolic BP > 85 mm or systolic BP >135 mm Hg after 5-10 minutes rest
* Body mass index (BMI) > 30.0 (or ≤18)
* Smoking in women who will be 35 years during the course of the trial; women < 35 years who smoke greater than 15 cigarettes per day must be evaluated by the PI for inclusion based on risk factors that would increase their risk for CVD and thromboembolism, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age.
* Women with severe cystoceles or rectoceles
* Use within the past 2 months of any implanted hormonal contraceptives including Mirena [progestin containing intrauterine system (IUS)] or Norplant (subdermal implant delivering LNG). NOTE: Removal of implanted hormonal contraceptives must have been for personal reasons unrelated to the purpose of enrollment in this study.
* Current use of a non-hormone containing IUD. NOTE: Removal of an IUD must have been for personal reasons unrelated to the purpose of enrollment in this study.
* Use of injectable contraceptives during the previous 3 months (e.g. Cyclofem) or 6 months (e.g. DMPA).
* Women who do not have at least two progesterone measurements during the control cycle of ≥10nmol/L will be excluded from further participation in the study (See Section 13.4.1)

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic efficacy as measured by the effects of a vaginal ring delivering Ulipristal acetate consistently combined with levonorgestrel administration on the endometrium | 3 months
  Endometrial biopsies (EB) will be taken as follows, a.During the follicular phase (between Day 9 and Day 12) of the baseline/control cycle, b. At the end of the 14th week of treatment (14 days after the 12 week LNG administration and end of CVR use), c. During the follicular phase (between Day 9 and Day 12 of the second menstrual cycle after ring removal). Also, endometrial changes will be measured by histological examination, immunohistochemistry, and assessment of proliferation markers (Ki67, Phospho H3 and bcl2).

SECONDARY OUTCOMES:
Safety as measured by number of participants with occurrence of adverse events (AEs) and concomitant medication use | 3 months
  Safety as measured by the assessment of a vaginal ring delivering Ulipristal acetate consistently combined with levonorgestrel administration

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Merkatz, Ph.D., Study Director — Population Council
Locations (1):
- Profamilia, Santo Domingo, Dominican Republic